CLINICAL TRIAL: NCT01556633
Title: An Open Label, Prospective, Single Oral Dose Study Evaluating the Pharmacokinetics, Safety, and Tolerability of Oseltamivir in Adult Subjects on Peritoneal Dialysis (PD) Using a Rapid Cycle Regimen to Simulate APD and in Adult Subjects With Creatinine Clearance From 10 to 30 mL/Min Not on Dialysis
Brief Title: A Single Dose Study of Tamiflu in Volunteers in Dialysis And in Volunteers With Reduced Creatinine Clearance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NV25655
Record Dates: First submitted 2012-03-15; First posted 2012-03-16 (Estimated); Results first posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Oseltamivir

ARMS (2):
- Volunteers on dialysis (Experimental)
  Interventions: Drug: Tamiflu (oseltamivir)
- Volunteers with reduced creatinine clearance (Experimental)
  Interventions: Drug: Tamiflu (oseltamivir)

INTERVENTIONS:
Drug: Tamiflu (oseltamivir) — Single dose of Tamiflu in volunteers on dialysis
  Arms: Volunteers on dialysis
Drug: Tamiflu (oseltamivir) — Single dose of Tamiflu in volunteers with creatinine clearance from 10 to 30 mL/min
  Arms: Volunteers with reduced creatinine clearance

SUMMARY:
This open-label, prospective, single dose study will evaluate the pharmacokinetics and safety of Tamiflu (oseltamivir) in volunteers on dialysis and in volunteers with a creatinine clearance from 10 to 30 mL/min. Volunteers will receive a single oral dose of Tamiflu.

ELIGIBILITY:
Inclusion Criteria:

General

* Adult volunteers, aged 19 to 90 years
* Medically stable with no hospitalization for a significant disease in the 3 months before study start

Volunteers on dialysis

* A documented and well-established dialysis therapy

Volunteers with reduced creatinine clearance

* Creatinine clearance from 10 to 30 mL/min
* Stable renal function

Exclusion Criteria:

* Clinically significant and unstable disease (e.g., cardiac, hepatic, pulmonary)
* Medical history of concurrent medical condition that would compromise participation in the study
* Hypotensive episodes or symptoms of fainting, dizziness or lightheadedness in the 4 weeks before screening
* Uncontrolled hypotension or hypertension
* Infection with hepatitis B, hepatitis C or human immunodeficiency virus

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- New Zealand (2):
  - Christchurch
  - Grafton

REFERENCES:
- [Derived] Patel K, Rayner CR, Giraudon M, Kamal MA, Morcos PN, Robson R, Kirkpatrick CM. Pharmacokinetics and safety of oseltamivir in patients with end-stage renal disease treated with automated peritoneal dialysis. Br J Clin Pharmacol. 2015 Apr;79(4):624-35. doi: 10.1111/bcp.12526. PMID 25289522

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 27 participants were screened and 16 participants were enrolled in the study. The study was conducted from 09 March 2012 to 23 June 2012 at two study centers in New Zealand.
Groups:
- Dialysis (Oseltamivir 75 mg): Participants on Peritoneal Dialysis (PD) using a rapid cycle regimen to simulate Automated Peritoneal Dialysis (APD) received a single oral dose of oseltamivir 75 mg capsule.
- Reduced Creatinine Clearance (Oseltamivir 30 mg): Participants with creatinine clearance from 10 to 30 milliliter (mL)/minute (min) not on dialysis received a single oral dose of oseltamivir 30 mg capsule.
Period: Overall Study
Arm/Group | Dialysis (Oseltamivir 75 mg) | Reduced Creatinine Clearance (Oseltamivir 30 mg)
Started | 10 | 6
Completed | 10 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: All participants who received the study drug, whether prematurely withdrawn from the study or not, were included.
Groups:
- Reduced Creatinine Clearance (Oseltamivir 30 mg): Participants with creatinine clearance (CLCR) from 10 to 30 milliliter (mL)/minute (min) not on dialysis received a single oral dose of oseltamivir 30 mg capsule.
- Total: Total of all reporting groups
Arm/Group | Dialysis (Oseltamivir 75 mg) | Reduced Creatinine Clearance (Oseltamivir 30 mg) | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.8 (16.62) | 66.3 (9.95) | 57.9 (15.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Total Dialysate Clearance for Automated Peritoneal Dialysis (CLDAPD) of Oseltamivir and Oseltamivir Carboxylate for 75 mg Dose
Description: CLDAPD is the total dialysate clearance for automated peritoneal dialysis, attributable to both continuous cycler-assisted peritoneal dialysis (CCPD) and continuous ambulatory peritoneal dialysis (CAPD), which was calculated with the recovery method over the dense blood sampling collection interval from 0 to 48 hours post-dose.
  CLDAPD = the amount excreted into dialysate from 0 to 48 hours (Aed[0-48])/ plasma area under the concentration-time curve from time zero through 48 hours (AUC[0-48])
  CLDCCPD = mean of CLDCCPD from the 2 CCPD sessions, calculated as CLDCCPD = (Aed[0-8]/AUC[0-8] + Aed[24-32]/AUC[24-32]) / 2
  CLDCAPD = mean of CLDCAPD from the 3 CAPD sessions, calculated as CLDCAPD = (Aed[8-16]/AUC[8-16] + Aed[16-24]/AUC[16-24] + Aed[32-48]/AUC[32-48]) / 3
Time Frame: CCPD: pre-dose (0)-2.67, 2.67-5.33, 5.33-8; CAPD: 8-16, 16-24; CCPD: 24-26.67, 26.67-29.33, 29.33-32; CAPD: 32-40, 40-48 hrs post-dose for urine; CCPD and CAPD:0.5, 1.33, 2, 2.5, 3, 4, 5, 6.67, 8, 10, 12, 14, 16, 20, 24, 28, 32, 48 hrs post-dose for blood
Population: Pharmacokinetic (PK) population: Only 9 participants were included for this analysis as they did not significantly violate the inclusion or exclusion criteria, deviate significantly from the protocol or if data was unavailable or incomplete which influence the PK analysis were excluded from the PK analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre (L)/hour (h)
Groups:
- Dialysis (Oseltamivir 75 mg): Participants on Peritoneal Dialysis using a rapid cycle regimen to simulate Automated Peritoneal Dialysis (APD) received a single oral dose of oseltamivir 75 mg capsule.
Arm/Group | Dialysis (Oseltamivir 75 mg)
Number analyzed (Participants) | 9
Litre (L)/hour (h)
  Oseltamivir, CLDAPD | NA (NA) — CLDAPD is a derived from CLDCCPD and CLDCAPD. Since CLDCAPD could not be calculated as no oseltamivir concentration was found in the dialysate; therefore, CLDAPD could not be derived.
  Oseltamivir, CLDCAPD | NA (NA) — CLDCAPD could not be calculated as no oseltamivir concentration was found in the dialysate.
  Oseltamivir, CLDCCPD | 0.183 (23.8)
  Oseltamivir Carboxylate CLDAPD | 0.230 (13.1)
  Oseltamivir Carboxylate, CLDCAPD | 0.187 (11.8)
  Oseltamivir Carboxylate, CLDCCPD | 0.326 (18.5)

2. Secondary Outcome: Number of Participants With Any Adverse Event (AEs) and Any Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with the intervention. An SAE is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect.
Time Frame: Approximately 7 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Dialysis (Oseltamivir 75 mg) | Reduced Creatinine Clearance (Oseltamivir 30 mg)
Number analyzed (Participants) | 10 | 6
participants
  Any AEs | 9 | 2
  Any SAEs | 1 | 0

3. Primary Outcome: AUC120, AUC168 and AUCinf of Oseltamivir and Oseltamivir Carboxylate for 75 mg Dose
Description: AUC120 is defined as the area under the plasma concentration-time curve from time zero through 120 hours post-dose, AUC168 is defined as the area under the plasma concentration-time curve from time zero through 168 hours post-dose, and AUCinf is defined as the area under the plasma concentration-time curve from time zero extrapolated to infinity. Oseltamivir carboxylate is a clinically active metabolite of oseltamivir.
Time Frame: Pre-dose; 0.5, 1.33, 2, 2.5, 3, 4, 5, 6.67, 8, 10, 12, 14, 16, 20, 24, 28, 32, 48, 72, 96, 120, 144, and 168 hrs post-dose
Population: PK population was used for this outcome measure. Only 9 participants were included, who did not significantly violate the inclusion/exclusion criteria, deviate significantly from protocol or with unavailable or incomplete data which influence PK analysis. Numbers of participants analyzed for the indicated drug/metabolite were denoted by "n".
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)*h/ milliliter (mL)
Arm/Group | Dialysis (Oseltamivir 75 mg)
Number analyzed (Participants) | 9
nanogram (ng)*h/ milliliter (mL)
  AUC120 oseltamivir (n = 6) | 175 (33.3)
  AUC168 oseltamivir (n = 6) | 175 (33.3)
  AUCinf oseltamivir (n = 6) | 175 (33.3)
  AUC120 oseltamivir carboxylate (n = 9) | 83400 (88.9)
  AUC168 oseltamivir carboxylate (n = 9) | 89200 (96.0)
  AUCinf oseltamivir carboxylate (n = 9) | 93800 (102.5)

4. Primary Outcome: AUCinf of Oseltamivir and Oseltamivir Carboxylate for 30 mg Dose
Description: AUCinf is defined as the area under the plasma concentration-time curve from time zero extrapolated to infinity. Oseltamivir carboxylate is a clinically active metabolite of oseltamivir.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Reduced Creatinine Clearance (Oseltamivir 30 mg)
Number analyzed (Participants) | 6
ng*h/mL
  AUCinf, oseltamivir (n = 3) | 64.7 (46.2)
  AUCinf, oseltamivir carboxylate (n = 6) | 8630 (56.3)

5. Primary Outcome: Cmax of Oseltamivir and Oseltamivir Carboxylate
Description: The Plasma Concentration (Cmax) is defined as maximum observed analyte concentration. Oseltamivir carboxylate is a clinically active metabolite of oseltamivir.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dialysis (Oseltamivir 75 mg) | Reduced Creatinine Clearance (Oseltamivir 30 mg)
Number analyzed (Participants) | 9 | 6
ng/mL
  Oseltamivir (n = 9,5) | 67.1 (79.4) | 22.1 (38.2)
  Oseltamivir carboxylate (n = 9,6) | 1710 (31.0) | 361 (27.4)

6. Primary Outcome: C120h, C168h and Clast of Oseltamivir and Oseltamivir Carboxylate for 75 mg Dose
Description: C120h is defined as the plasma concentration at 120 hours post-dose. C168h is defined as the plasma concentration at 168 hours post-dose. Clast is defined as the plasma concentration corresponding to the time of the last measureable (positive) plasma concentration.
  Oseltamivir carboxylate is a clinically active metabolite of oseltamivir.
Time Frame: as for outcome 3
Population: PK population was used for this outcome measure. Only 9 participants were included, who did not significantly violate the inclusion/exclusion criteria, deviate significantly from protocol or with unavailable or incomplete data which influence PK analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dialysis (Oseltamivir 75 mg)
Number analyzed (Participants) | 9
ng/mL
  C120h, oseltamivir | NA (NA) — For all participants the oseltamivir concentration was below lower limit of quantification and therefore a mean could not be calculated.
  C168h,oseltamivir | NA (NA) — For all participants the oseltamivir concentration was below lower limit of quantification and therefore a mean could not be calculated.
  Clast, oseltamivir | 1.30 (0.271)
  C120h, oseltamivir carboxylate | 301.0 (264.0)
  C168h,oseltamivir carboxylate | 138.0 (135.0)
  Clast, oseltamivir carboxylate | 140.0 (132.0)

7. Primary Outcome: Tmax and T1/2 of Oseltamivir and Oseltamivir Carboxylate
Description: The Time of observed maximum plasma concentration (Tmax) is defined as actual sampling time to reach maximum observed analyte concentration.
  The Elimination Half-Life Period (T1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. Oseltamivir carboxylate is a clinically active metabolite of oseltamivir.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: h
Arm/Group | Dialysis (Oseltamivir 75 mg) | Reduced Creatinine Clearance (Oseltamivir 30 mg)
Number analyzed (Participants) | 9 | 6
h
  Tmax, Oseltamivir (n = 9, 5) | 2.50 [0.50 to 4.00] | 1.33 [0.50 to 4.00]
  T1/2, Oseltamivir (n = 6,3) | 1.92 [1.01 to 2.41] | 2.25 [1.12 to 3.39]
  Tmax, Oseltamivir carboxylate (n = 9, 6) | 20.00 [6.67 to 28.00] | 7.34 [6.67 to 12.07]
  T1/2, Oseltamivir Carboxylate (n = 9,6) | 35.3 [10.0 to 47.3] | 10.7 [8.87 to 21.0]

8. Primary Outcome: Renal Clearance (CLR) of Oseltamivir and Oseltamivir Carboxylate
Description: CLR is calculated as the cumulative amount of drug excreted into urine from 0 to time t hours (Ae0-tlast) / area under the concentration-time curve from time zero through the last quantifiable concentration time (AUC0-t).
Time Frame: Pre-dose; 0.5, 1.33, 2, 2.5, 3, 4, 5, 6.67, 8, 10, 12, 14, 16, 20, 24, 28, 32, 48, 72, 96, 120, 144, and 168 hrs post-dose for blood; pre-dose and 0-24, 24-48, 48-72, 72-96, 96-120, 120-144, and 144-168 hrs post-dose for urine.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Dialysis (Oseltamivir 75 mg) | Reduced Creatinine Clearance (Oseltamivir 30 mg)
Number analyzed (Participants) | 9 | 6
L/h
  CLR, oseltamivir (n = 4, 5) | 0.572 (441.3) | 3.30 (70.6)
  CLR, oseltamivir carboxylate (n = 4, 6) | 0.655 (217.4) | 2.28 (81.3)

9. Secondary Outcome: Number of Participants With Marked Abnormality in Laboratory Measurements
Description: Laboratory analysis included: hematology (hemoglobin, hematocrit, reticulocyte, red blood cell, platelet and white blood cell count, mean corpuscular volume, mean corpuscular hemoglobin), prothrombin and activated partial thromboplastin time, biochemistry (sodium, potassium, bicarbonate, phosphate, chloride, calcium, urea, serum creatinine, bilirubin, cholesterol, alkaline phosphatase, aspartate aminotransferase, alanine aminotransferase [ALT], gamma-glutamyl transferase, protein, albumin, amylase, creatinine, lipase), random glucose, and urinalysis.
  Laboratory test result values falling outside of the marked abnormality range that also represent a defined change from baseline were considered as marked laboratory abnormalities. A marked reference range for sodium is 130-150 millimole (mmol)/L, chloride is 95-115 mmol/L, phosphate is 0.75-1.60 mmol/L, calcium is 2-2.90 mmol/L, glucose is 2.8-11.10 mmol/L, bicarbonate is 18-28 mmol/L, and ALT is 0-110 Unit/L.
Time Frame: Approximately 7 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Dialysis (Oseltamivir 75 mg) | Reduced Creatinine Clearance (Oseltamivir 30 mg)
Number analyzed (Participants) | 10 | 6
participants
  Sodium chloride | 1 | 0
  Chloride | 3 | 0
  Phosphate | 3 | 0
  Calcium | 1 | 0
  Glucose (random) | 1 | 0
  Bicarbonate | 1 | 0
  ALT | 1 | 0

10. Secondary Outcome: Number of Participants With Change From Baseline in Marked Abnormality in Electrocardiogram (ECG) Parameters at Follow-up Visit
Description: ECG parameter included QT interval, QTcB interval and QTcF interval (all intervals are measured in millisecond [msec]). Marked abnormality in ECG is predefined for QT, QTcB, and QTcF interval as <=30, >30-60, and >60 msec increase from baseline.
Time Frame: From Baseline (Day -1) to Follow-up visit (Days 15 to 22)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Dialysis (Oseltamivir 75 mg) | Reduced Creatinine Clearance (Oseltamivir 30 mg)
Number analyzed (Participants) | 10 | 6
participants
  QT, <= 30 | 8 | 6
  QT, > 30 - 60 | 2 | 0
  QTcB, <= 30 | 10 | 6
  QTcF, <= 30 | 9 | 6
  QTcF, > 30 - 60 | 1 | 0

11. Secondary Outcome: Number of Participants With Abnormal Shifts in Vital Signs
Description: Vital signs included pulse rate, systolic blood pressure (SBP), diastolic blood pressure (DBP), and body temperature.
  Vital sign with abnormal shifts from normal at baseline to high or low at post-baseline time points were recorded. Blood pressure was recorded in millimeter of mercury (mmHg), and temperature in degrees Celsius. Low blood pressure defined as <=70 mmHg (SBP) and <=40 mmHg (DBP); high blood pressure defined as >=140 mmHg (SBP) and >=90 mmHg (DBP); low temperature defined as <=36.5 degrees Celsius and high temperature defined as >=37.5 degrees Celsius.
Time Frame: Days 1 (post-dose), 2, 3, 4, 5, 6, 7, 8; and Follow-up visit (Days 15 to 22)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Dialysis (Oseltamivir 75 mg) | Reduced Creatinine Clearance (Oseltamivir 30 mg)
Number analyzed (Participants) | 10 | 6
participants
  SBP , Day 1 - postdose, High | 1 | 0
  SBP, Day 2, High | 2 | 1
  SBP, Day 3, High | 2 | 1
  SBP, Day 4, High | 2 | 1
  SBP, Day 5, High | 2 | 1
  SBP, Day 7, High | 1 | 1
  SBP, Day 8, High | 1 | 0
  SBP, Follow Up, High | 2 | 0
  DBP, Day 2, High | 0 | 1
  DBP, Day 3, High | 2 | 0
  DBP, Day 7, High | 0 | 1
  DBP, Day 8, High | 0 | 1
  DBP, Follow Up, High | 3 | 0
  Temperature, Day 4, Low | 2 | 0
  Temperature, Day 6, Low | 1 | 0
  Temperature, Day 7, Low | 1 | 0
  Temperature, Day 8, Low | 1 | 0
  Temperature, Follow Up, Low | 2 | 0

ADVERSE EVENTS:
Time Frame: Approximately 7 weeks
Description: Safety population: All participants who received the study drug, whether prematurely withdrawn from the study or not, were included.
Arm/Group | Dialysis (Oseltamivir 75 mg) | Reduced Creatinine Clearance (Oseltamivir 30 mg)
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/6
Other Adverse Events (participants affected / at risk) | 9/10 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dialysis (Oseltamivir 75 mg) (N=10) | Reduced Creatinine Clearance (Oseltamivir 30 mg) (N=6)
Respiratory tract infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dialysis (Oseltamivir 75 mg) (N=10) | Reduced Creatinine Clearance (Oseltamivir 30 mg) (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Infrequent bowel movements (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Catheter site hematoma (General disorders) | 1 | 0
Edema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dizziness postural (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Lethargy (Nervous system disorders) | 1 | 0
Parasthesia (Nervous system disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.